CLINICAL TRIAL: NCT05304793
Title: A Pilot Study to Test a Cognitive-Behavioral Model for Dyspnea in Patients With Lung Cancer
Brief Title: Testing a Cognitive Behavioral Model for Reducing Dyspnea in Patients With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Barbara Andersen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-20089; NCI-2020-08108 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-03-03; First posted 2022-03-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Lung Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Practice Guidelines as Topic; Standard of Care; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (TAB) (Experimental): Patients participate in 4 weekly TAB in-person or video conference sessions over 1 hour each that provide them with skills to cope with their dyspnea. Patients also receive treatment handouts, a CD with an audio file with instructions for progressive muscle relaxation, and a pulse oximeter. Patients may receive additional support calls over 10-15 minutes from the TAB provider within 1 week following each session.
  Interventions: Behavioral: Cognitive Behavior Therapy; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patients receive usual management of dyspnea from the treating physician.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual management of dyspnea
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Behavioral: Cognitive Behavior Therapy — Receive TAB treatment
  Other Names: CBT; cognitive therapy; CT
  Arms: Arm I (TAB)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the effect of a form of cognitive-behavioral therapy, Take a Breath, on reducing the intensity and frequency of dyspnea (difficulty breathing) in patients with lung cancer. Take a Breath consists of individual therapy sessions that educate patients on dyspnea and provides coping strategies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the acceptability (based on patient satisfaction), tolerability (based on rate of symptom exacerbation from pre- to post-treatment), and feasibility (based on number of patients agreeing to be participate, adherence rate, and retention rate of treatment) of Take a Breath (TAB), a skills-based cognitive-behavioral treatment lasting 4 weekly hour-long sessions targeting dyspnea and related distress and impairment, in adults with lung cancer (N=40).

SECONDARY OBJECTIVES:

I. To provide preliminary data on the effectiveness of TAB on dyspnea and related distress and impairment.

II. To test cognitive-behavioral variables (physical symptoms, thoughts, behaviors, and emotions) as predictors of dyspnea severity and anxiety sensitivity as a moderator.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients participate in 4 weekly TAB in-person or video conference sessions over 1 hour each that provide them with skills to cope with their dyspnea. Patients also receive treatment handouts, a compact disk (CD) with an audio file with instructions for progressive muscle relaxation, and a pulse oximeter. Patients may receive additional support calls over 10-15 minutes from the TAB provider within 1 week following each session.

ARM II: Patients receive usual management of dyspnea from the treating physician.

After completion of study, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC)
* Currently experiencing dyspnea as defined by a score >= 1 on the American Thoracic Society (ATS) Dyspnea Questionnaire within 3 weeks of enrollment
* Seeking medical oncology care and treatment at the Ohio State University Comprehensive Cancer Center (OSUCCC) Thoracic Oncology Clinic
* Ability to understand and willingness to sign an informed consent document

Exclusion Criteria:

* Presence of other serious comorbidities that would interfere with patients' study participation (e.g., serious mental illness, heart disease) as determined by the treating oncologist
* Life expectancy < 2 months
* History of surgery for lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Change in acceptability of Take a Breath (TAB) | Baseline up to 1 month post-treatment
  Will be based on patient satisfaction scores using the Client Satisfaction Questionnaire, and will be determined to be acceptable if patient satisfaction scores at least "moderately" satisfied. To determine change over time in TAB, each analysis will include: covariates selected based on significant spearman correlation with outcomes, time (fixed), and time (random). To determine a differential rate of change in outcomes between TAB and treatment as usual (TAU), each analysis will include: covariates selected based on significant spearman correlation with outcomes, time (fixed), time (random), condition (fixed) and the fixed interaction between time and condition (time x condition).
Change in tolerability of TAB | Baseline up to 1 month post-treatment
  Will be based on the change in dyspnea symptoms from pre- to post-treatment, and determined to be tolerable if there is not a significant increase in dyspnea symptoms at post-treatment. To determine change over time in TAB, each analysis will include: covariates selected based on significant spearman correlation with outcomes, time (fixed), and time (random). To determine a differential rate of change in outcomes between TAB and TAU, each analysis will include: covariates selected based on significant spearman correlation with outcomes, time (fixed), time (random), condition (fixed) and the fixed interaction between time and condition (time x condition).
Feasibility of TAB | Up to 1 month post-treatment
  Based on patient enrollment (% of eligible patients enrolled to the study) and treatment adherence (% of patients retained in the study)
Change in dyspnea severity using the American Thoracic Society Dyspnea Questionnaire | Baseline up to 1 month post-treatment
  Will be assessed per the American Thoracic Society (ATS) Dyspnea Questionnaire. The ATS Dyspnea Questionnaire is a 5-item self-report measure of dyspnea with higher scores indicating greater severity. This scale was developed for epidemiological research and is a common, brief clinical measure of dyspnea. Items are summed with scores ranging from 0-5. Responses of 0 indicate no dyspnea while responses ≥1 indicate experiences of dyspnea.
Change in shortness of breath | Baseline up to 1 month post-treatment
  Will be assessed per the Shortness of Breath Questionnaire. The BCS is a 13-item self-report measure of catastrophic thoughts regarding breathlessness[59]. Patients rate "the degree to which you have these thoughts and feelings when you are experiencing breathlessness" (e.g., "I feel I can't go on"). Each item is rated on a 5-point Likert scale (0=not at all to 4=all the time). The BCS is a reliable measure and was originally validated in patients with severe COPD.

SECONDARY OUTCOMES:
Mood disturbance | Up to 1 month post-treatment
  The POMS-SF is a 37-item self-report measure of psychological distress. Patients are asked to indicate the degree to which each item, a moodrelated adjective (e.g., tense), describes themselves on a 5-point Likert scale (0=not at all to 4=extremely). The POMS-SF provides an overall Total Mood Disturbance score as well as scores for each of the six subscales (tension-anxiety, depression, anger-hostility, vigor-activity, fatigue, and confusion-bewilderment)
Catastrophic thoughts related to dyspnea | Up to 1 month post-treatment
  e BCS is a 13-item self-report measure of catastrophic thoughts regarding breathlessness[59]. Patients rate "the degree to which you have these thoughts and feelings when you are experiencing breathlessness" (e.g., "I feel I can't go on"). Each item is rated on a 5-point Likert scale (0=not at all to 4=all the time). The BCS is a reliable measure and was originally validated in patients with severe COPD.
Physical activity using International Physical Activity Questionnaire (IPAQ) | Up to 1 month post-treatment
  The IPAQ is a 7-item measure of physical activity conducted over the previous week. Participants are asked to list the amount of time they engaged in each of the listed activities (e.g. During the last 7 days, how much time did you spend sitting on a week day?). Extensive reliability and validity testing undertaken across 12 countries indicates that this measure demonstrates strong psychometric properties

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Andersen, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo SB, Arrato NA, Presley CJ, McGinty HL, Otto MW, Andersen BL. Cognitive-Behavioral Treatment for Breathlessness in Lung Cancer: A Randomized Controlled Trial. Ann Am Thorac Soc. 2025 Oct;22(10):1579-1591. doi: 10.1513/AnnalsATS.202406-580OC. PMID 40772929
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05304793/ICF_000.pdf